CLINICAL TRIAL: NCT05328908
Title: A Phase 3, Randomized, Open-label Study of Relatlimab-nivolumab Fixed-dose Combination Versus Regorafenib or Trifluridine + Tipiracil (TAS-102) for Participants With Later-lines of Metastatic Colorectal Cancer
Brief Title: A Study of Nivolumab-relatlimab Fixed-dose Combination Versus Regorafenib or TAS-102 in Participants With Later-lines of Metastatic Colorectal Cancer
Acronym: RELATIVITY-123
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability to meet protocol objectives
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-123; 2021-004285-35 (EudraCT Number)
Expanded Access: NCT05170685 (No longer available)
Record Dates: First submitted 2022-03-14; First posted 2022-04-14 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Neoplasms
Keywords: Micro-satellite Stable (MSS) Metastatic Colorectal Cancer (mCRC); Relatlimab; Nivolumab; BMS-986213; Regorafenib; Stivarga; Lonsurf
MeSH Terms: conditions — Colorectal Neoplasms; Spinocerebellar Degenerations | interventions — regorafenib; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab + Relatlimab Fixed-dose Combination (FDC) (Experimental)
  Interventions: Drug: Nivolumab-relatlimab FDC
- Arm B: Investigator's Choice (Active Comparator): Treatment with Regorafenib or TAS-102
  Interventions: Drug: Regorafenib; Drug: TAS-102

INTERVENTIONS:
Drug: Nivolumab-relatlimab FDC — Specified dose on specified days
  Other Names: BMS-986213
  Arms: Arm A: Nivolumab + Relatlimab Fixed-dose Combination (FDC)
Drug: Regorafenib — Specified dose on specified days
  Other Names: Stivarga
  Arms: Arm B: Investigator's Choice
Drug: TAS-102 — Specified dose on specified days
  Other Names: Trifluridine/Tipiracil; Lonsurf
  Arms: Arm B: Investigator's Choice

SUMMARY:
The purpose of this study is to evaluate relatlimab in combination with nivolumab, administered as a fixed-dose combination (nivolumab-relatlimab FDC, also referred to as BMS-986213) for the treatment of non-microsatellite instability high (MSI-H)/deficient mismatch repair (dMMR) metastatic colorectal cancer (mCRC) participants who failed at least 1 but no more than 4 prior lines of therapy for metastatic disease.

ELIGIBILITY:
Inclusion Criteria

* Histological confirmed previously treated colorectal cancer with adenocarcinoma histology with metastatic or recurrent unresectable disease at study entry.
* Participants must have:.

  i) progressed during or within approximately 3 months following the last administration of approved standard therapies (at least 1, but not more than 4 prior lines of therapies in the metastatic setting), which must include a fluoropyrimidine, oxaliplatin, irinotecan, an anti-VEGF therapy, and anti-EGFR therapy (if RAS wild-type), if available in the respective country, or;.

ii) been intolerant to prior systemic chemotherapy regimens if there is documented evidence of clinically significant intolerance despite adequate supportive measures.

* Must have sufficient tumor tissue & evaluable PD-L1 expression to meet the study requirements.
* Must have measurable disease per RECIST v1.1. Participants with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll provided the lesion(s) have demonstrated clear progression and can be measured accurately.

Exclusion Criteria

* Prior treatment with either an immunotherapy or with regorafenib or with TAS-102.
* Untreated central nervous system (CNS) metastases, participants are eligible if CNS metastases have been treated and participants have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment).
* History of refractory hypertension not controlled with anti-hypertensive therapy, myocarditis (regardless of etiology), uncontrolled arrhythmias, acute coronary syndrome within 6 months prior to dosing, Class II congestive heart failure (as per the New York Heart Association Functional Classification), interstitial lung disease/pneumonitis or an active, known or suspected autoimmune disease.
* Confirmed tumor microsatellite instable high/deficient mismatch repair (MSI-H/dMMR) status as per local standard testing; MSI/MMR test results from initial diagnosis are acceptable.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) in randomized participants with programmed death-ligand 1 (PD-L1) combined positive score (CPS) ≥ 1 | Up to 5 years after last participant randomized
OS in all randomized participants | Up to 5 years after last participant randomized

SECONDARY OUTCOMES:
Objective response rate (ORR) by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 in randomized participants with PD-L1 CPS ≥ 1 | Up to 5 years after last participant randomized
ORR by BICR per RECIST v1.1 in all randomized participants | Up to 5 years after last participant randomized
Progression-free survival (PFS) by BICR per RECIST v1.1 in randomized participants with PD-L1 CPS ≥ 1 | Up to 5 years after last participant randomized
PFS by BICR per RECIST v1.1 in all randomized participants | Up to 5 years after last participant randomized
Duration of response (DoR) by BICR per RECIST v1.1 in responders with PD-L1 CPS ≥ 1 | Up to 5 years after last participant randomized
DoR by BICR per RECIST v1.1 in all responders | Up to 5 years after last participant randomized
Number of participants with adverse events (AEs) | Up to 135 days after participant's last dose
Number of participants with serious adverse events (SAEs) | Up to 135 days after participant's last dose
Number of participants with immune-mediated adverse events (IMAEs) | Up to 135 days after participant's last dose
Number of participants with AEs leading to discontinuation | Up to 135 day's after participant's last dose
Number of participants with clinical laboratory abnormalities | Up to 135 days after participant's last dose
Time Until Definitive Deterioration-Physical Function (TUDD-PF): The time from randomization until definitive deterioration in the EORTC QLQ-C30 physical function scale score in randomized participants with PD-L1 CPS ≥ 1 | Up to follow up visit 2 (approximately 135 days after last dose)
  The EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire-Core 30 (QLQ-C30) consists of 30 questions incorporated into 5 functional scales (physical, role, cognitive, emotional, and social functioning), 3 multi-item symptom scales (fatigue, pain, nausea and vomiting), a global health status / Quality of Life scale, and six single symptom items. All of the scale and single-item measures range in score from 0 to 100, where a higher score represents a higher response level. High functional scores indicates more favorable outcomes and a higher score on the symptom domains indicates higher symptom burden/less favorable patient outcome.
TUDD-PF: The time from randomization until definitive deterioration in the EORTC QLQ-C30 physical function scale score in all randomized participants | Up to follow up visit 2 (approximately 135 days after last dose)
TUDD-QoL: The time from randomization until definitive deterioration in the EORTC QLQ-C30 global health status/QoL scale score in randomized participants with PD-L1 CPS ≥ 1 | Up to follow up visit 2 (approximately 135 days after last dose)
  QoL = Quality of Life. The EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire-Core 30 (QLQ-C30) consists of 30 questions incorporated into 5 functional scales (physical, role, cognitive, emotional, and social functioning), 3 multi-item symptom scales (fatigue, pain, nausea and vomiting), a global health status / Quality of Life scale, and six single symptom items. All of the scale and single-item measures range in score from 0 to 100, where a higher score represents a higher response level. High functional scores indicates more favorable outcomes and a higher score on the symptom domains indicates higher symptom burden/less favorable patient outcome.
TUDD-QoL: The time from randomization until definitive deterioration in the EORTC QLQ-C30 global health status/QoL scale score in all randomized participants | Up to follow up visit 2 (approximately 135 days after last dose)
PFS by investigator per RECIST v1.1 in randomized participants with PD-L1 CPS ≥ 1 | Up to 5 years after last participant randomized
PFS by investigator per RECIST v1.1 in all randomized participants | Up to 5 years after last participant randomized
ORR by investigator per RECIST v1.1 in randomized participants with PD-L1 CPS ≥ 1 | Up to 5 years after last participant randomized
ORR by investigator per RECIST v1.1 in all randomized participants | Up to 5 years after last participant randomized
DoR by investigator per RECIST v1.1 in responders with PD-L1 CPS ≥ 1 | Up to 5 years after last participant randomized
DoR by investigator per RECIST v1.1 in all randomized participants | Up to 5 years after last participant randomized

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (139):
- United States (20):
  - Local Institution - 0044, Springdale, Arkansas
  - Local Institution - 0012, Los Angeles, California
  - Local Institution - 0117, Norwich, Connecticut
  - Local Institution - 0025, Miami, Florida
  - Local Institution - 0031, Atlanta, Georgia
  - Local Institution - 0071, Boise, Idaho
  - Local Institution - 0081, Fort Wayne, Indiana
  - Massachusetts General Hospital,, Boston, Massachusetts
  - Local Institution - 0042, Ann Arbor, Michigan
  - Local Institution - 0043, East Brunswick, New Jersey
  - Local Institution - 0009, Durham, North Carolina
  - Local Institution - 0082, Cincinnati, Ohio
  - Local Institution - 0095, Columbus, Ohio
  - Local Institution - 0147, Philadelphia, Pennsylvania
  - Local Institution - 0008, Charleston, South Carolina
  - Local Institution - 0096, Sioux Falls, South Dakota
  - Local Institution - 0127, Nashville, Tennessee
  - Local Institution - 0097, Fort Worth, Texas
  - Local Institution - 0132, Richmond, Virginia
  - Local Institution - 0005, Madison, Wisconsin
- Argentina (4):
  - Local Institution - 0022, Ciudad Autónoma Buenos Aires, Buenos Aires
  - Local Institution - 0026, Ciudad Autónoma Buenos Aires, B
  - Local Institution - 0024, Ciudad Autónoma Buenos Aires
  - Local Institution - 0023, Río Grande
- Australia (6):
  - Local Institution - 0098, Wagga Wagga, New South Wales
  - Local Institution - 0114, Westmead, New South Wales
  - Local Institution - 0001, Greenslopes, Queensland
  - Local Institution - 0010, Clayton, Victoria
  - Local Institution - 0021, Melbourne, Victoria
  - Local Institution - 0027, Murdoch, Western Australia
- Austria (3):
  - Local Institution - 0030, Graz
  - Local Institution - 0078, Klagenfurt
  - Local Institution - 0131, Salzburg
- Belgium (4):
  - Local Institution - 0062, Woluwé-Saint-Lambert, BRU
  - Local Institution - 0068, Ghent, VOV
  - Local Institution - 0070, Edegem
  - Local Institution - 0120, Leuven
- Canada (6):
  - Local Institution - 0003, Edmonton, Alberta
  - Local Institution - 0014, Ottawa, Ontario
  - Local Institution - 0007, Toronto, Ontario
  - Local Institution - 0019, Montreal, Quebec
  - Local Institution - 0104, Montreal, Quebec
  - Local Institution - 0004, Sherbrooke, Quebec
- Chile (2):
  - Local Institution - 0015, Santiago, RM
  - Local Institution - 0033, Santiago, RM
- China (18):
  - Local Institution - 0134, Chongqing, CQ
  - Local Institution - 0151, Guangzhou, Guangdong
  - Local Institution - 0126, Wuhan, HB
  - Local Institution - 0138, Changsha, HN
  - Local Institution - 0164, Wuhan, Hubei
  - Local Institution - 0158, Changsha, Hunan
  - Local Institution - 0146, Huaian, Jiangsu
  - Local Institution - 0143, Nanjing, JS
  - Local Institution - 0142, Jinan, SD
  - Local Institution - 0152, Xi'an, SHA
  - Local Institution - 0144, Chengdu, Sichuan
  - Local Institution - 0141, Taiyuan, SX
  - Local Institution - 0150, Tianjin, TJ
  - Local Institution - 0160, Hangzhou, ZJ
  - Local Institution - 0122, Beijing
  - Local Institution - 0139, Hangzhou
  - Local Institution - 0153, Shanghai
  - Local Institution - 0149, Shenyang
- Czechia (5):
  - Local Institution - 0099, Hořovice
  - Local Institution - 0016, Hradec Králové
  - Local Institution - 0100, Olomouc
  - Local Institution - 0123, Ostrava
  - Local Institution - 0064, Prague
- France (7):
  - Local Institution - 0066, Bordeaux
  - Local Institution - 0017, Caen
  - Local Institution - 0090, Dijon
  - Local Institution - 0020, Levallois-Perret
  - Local Institution - 0036, Lyon
  - Local Institution - 0089, Paris
  - Local Institution - 0039, Suresnes
- Germany (8):
  - Local Institution - 0054, Mannheim, Baden-Wurttemberg
  - Local Institution - 0056, Reutlingen, Baden-Wurttemberg
  - Local Institution - 0053, Würzburg, Bavaria
  - Local Institution - 0041, Frankfurt A. Main, Hesse
  - Local Institution - 0101, Essen, Northwest
  - Local Institution - 0055, Berlin, State of Berlin
  - Local Institution - 0040, Hamburg
  - Local Institution - 0034, München
- Italy (8):
  - Local Institution - 0046, Milan, MI
  - Local Institution - 0148, Padua, PD
  - Local Institution - 0059, Reggio Emilia, RE
  - Local Institution - 0060, Catania
  - Local Institution - 0091, Genova
  - Local Institution - 0045, Milan
  - Local Institution - 0115, Napoli
  - Local Institution - 0061, Napoli
- Japan (14):
  - Local Institution - 0110, Osaka, Osaka
  - Local Institution - 0107, Chiba
  - Local Institution - 0103, Chūōku
  - Local Institution - 0105, Hidaka-shi
  - Local Institution - 0154, Kasama-Shi
  - Local Institution - 0084, Kashiwa-Shi
  - Local Institution - 0086, Kawasaki-Shi
  - Local Institution - 0119, Kitaadachi-gun
  - Local Institution - 0108, Kōtoku
  - Local Institution - 0118, Matsuyama
  - Local Institution - 0088, Sapporo
  - Local Institution - 0083, Suita-Shi
  - Local Institution - 0085, Sunto-gun
  - Local Institution - 0124, Yokohama
- Local Institution - 0050, Amsterdam, Netherlands
- Poland (4):
  - Local Institution - 0051, Warsaw, Masovian Voivodeship
  - Local Institution - 0037, Warsaw, Pl-mz
  - Local Institution - 0018, Krakow
  - Local Institution - 0052, Warsaw
- Local Institution - 0106, San Juan, PR, Puerto Rico
- Singapore (2):
  - Local Institution - 0109, Singapore
  - Local Institution - 0087, Singapore
- South Korea (6):
  - Local Institution - 0072, Seoul, Seoul-teukbyeolsi
  - Local Institution - 0073, Goyang-si, Gyeonggi-do
  - Local Institution - 0129, Seongnamsi Bundanggu
  - Local Institution - 0092, Seoul
  - Local Institution - 0075, Seoul
  - Local Institution - 0074, Seoul
- Spain (8):
  - Local Institution - 0029, Badalona, B
  - Local Institution - 0093, Barcelona, B
  - Local Institution - 0102, Madrid, M
  - Local Institution - 0116, Zaragoza, Z
  - Local Institution - 0112, A Coruña
  - Local Institution - 0080, Barcelona
  - Local Institution - 0113, Madrid
  - Local Institution - 0035, Seville
- Sweden (5):
  - Local Institution - 0038, Stockholm, AB
  - Local Institution - 0135, Stockholm, AB
  - Local Institution - 0058, Uppsala, C
  - Local Institution - 0067, Gothenburg
  - Local Institution - 0094, Malmo
- Switzerland (2):
  - Local Institution - 0057, Aarau, Canton of Aargau
  - Local Institution - 0069, Bern
- Taiwan (5):
  - Local Institution - 0128, Changhua, CHA
  - Local Institution - 0111, Kaohsiung City, KHH
  - Local Institution - 0076, Tainan, TNN
  - Local Institution - 0121, Zhongzheng, TPE
  - Local Institution - 0077, Tainan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com